CLINICAL TRIAL: NCT06581549
Title: From Immune Microenvironment Characterization and Gene Expression Profiling to New Drugs Testing in Pleural and Peritoneal Mesothelioma: Imaging-Meso Study
Brief Title: Immune Microenvironment and Gene Expression Profiling in Mesothelioma
Acronym: Imaging-Meso
Status: Recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Imaging-Meso study
Record Dates: First submitted 2024-08-07; First posted 2024-09-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Mesothelioma; Mesotheliomas Pleural; Mesothelioma; Lung
Keywords: pleura; mesothelioma; PPM patients; lung; Gene expression profiling; Immune microenvironment
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Translation analysis — Bulk GEP analysis, Spatial whole transcriptome analysis, mIF analysis of tumors

SUMMARY:
Pleural and peritoneal mesotheliomas (PPM) are rare cancers mostly related to asbestos-exposure, which are characterized by a complex histopathological diagnosis and staging, few therapeutic options and a dismal prognosis. The main unmet medical need in PPM is the lack of a treatment sequence for affected patients. The advent of immune checkpoint inhibitors has changed the first line treatment of PPM, thanks to the improvement in survival achieved by the combination of ipilimumab and nivolumab that are currently approved for non-epithelioid histology in our Country.

PPM is characterized by a large heterogeneity of the genomic landscape, which is mainly characterized by the loss of tumour suppressor genes and mutations in DNA repair genes and by an "altered- suppressed" or "excluded" tumor immune microenvironment (TIME).

The goal of this project is to improve the immune-biological and molecular stratification of PPM subgroups that can lead to the identification of different personalized treatment approaches. PPM patients (N=220) will be retrospectively (N=150) and prospectively (N=70) recruited from the coordinator center and 6 participating Italian centers. Treatment-naïve tumor samples will be collected and analyzed by bulk gene expression and spatial whole transcriptome analysis, and by 9-color multiplex immunofluorescence.

New targets or actionable pathways potentially emerging from such studies will be finally assessed and validated in patient-derived organoids/xenografts that accurately reflect PPM tumorigenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Mesothelioma of the Pleura and Peritoneum
* Age greater than 18 years of age
* Patients undergoing surgery will require both biopsy and surgical sampling material
* Pathologist's confirmation of the presence of tumor sections in the excised specimens
* Patients in follow-up from active cancer treatment for at least 6 months

Exclusion Criteria:

* Inadequacy of biological material for analysis under study
* Patients not amenable to active oncologic treatment
* Patients lost to follow-up before 6 months after the end of active oncologic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 220 PPM patients will be enrolled in 7 Centers, 150 retrospectively and 70 prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | Through study completion, an average of 3 years
  PPM treatment-naïve tumor samples and classification in different clusters according to the differential expression of molecular and gene signatures by Gene expression profile (GEP) analysis.
Primary outcome | Through study completion, an average of 3 years
  Identification of molecular and immune signatures predictive of resistance or sensitivity to systemic anticancer drugs: chemotherapy or immunotherapy administered as first line treatment by spatial whole transcriptome analysis.
Primary outcome | Through study completion, an average of 3 years
  PPM surgical specimens and comparison with GEP in matched treatment-naïve tumor samples will be performed by gene expression profile analysis with GEP analysis.

SECONDARY OUTCOMES:
Secondary outcome | Through study completion, an average of 3 years
  Characterization and quantification of immune cell distribution and their spatial relationships in treatment naïve tumor samples of PPM patients will be performed by a 9-color multiplex immunofluorescence (mIF) analysis.
Secondary outcome | Through study completion, an average of 3 years
  Immune phenotypes defined by mIF and the immune signatures identified by GEP analyses will be performed in each treatment-naïve tumor sample.

OTHER OUTCOMES:
Third outcome | Through study completion, an average of 3 years
  In vitro and in vivo models of PPM for the investigation of activated signatures, new therapeutic targets and drug sensitivity tests. will be performed by:
  * development of in vitro 'organ-like' 3D structures (PDOs) derived from patient tumor tissue;
  * patient-derived xenograft (PDX) from PPM patients;
  * matched comparison of histological and molecular features of PDOs and PDXs with the original tumor tissues;
  * drug sensitivity/resistance tests in vitro and in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Pasello, MD, Principal Investigator — Istituto Oncologico Veneto IOV IRCCS
Locations (10):
- Italy (10):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Centro di Riferimento Oncologico (CRO) IRCCS, Aviano, Pordenone
  - Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Asst Papa Giovanni Xxiii Bergamo, Bergamo
  - Ircss Ospedale Policlinico San Martino, Genova
  - Asst Grande Ospedale Metropolitano Niguarda-Milano, Milan
  - Fondazione Ircss Istituto Nazionale Dei Tumori Di Milano, Milan
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera-Universitaria di Parma, Parma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona

IPD SHARING:
Plan to Share IPD: No